CLINICAL TRIAL: NCT04570696
Title: Measurement of the Plasmatic TFPI Level in Haemophilia Patients and Correlation With Thrombin Generation Assay (TGA) Parameters
Brief Title: TFPI Levels in Haemophilia A and B Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO19085
Record Dates: First submitted 2020-09-23; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Haemophilia A and B
Keywords: Haemophilia; TFPI inhibitors; TGA; TFPI
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult haemophilia patients: Adult (≥ 18 years old) haemophilia patients, only men
  Interventions: Other: NON INTERVENTIONAL

INTERVENTIONS:
Other: NON INTERVENTIONAL — NON INTERVENTIONAL

SUMMARY:
The goal of this study is to measure the TFPI plasma level, a molecule involved in the regulation of the coagulation system, in haemophilia patients. The second objective is to assess the effects of TFPI inhibition on thrombin generation. Indeed, there is sparse data on the physiological and pathological changes of TFPI levels in human and particularly in hemophilia patients. Yet, TFPI inhibitors may become one of the new by-passing treatments of haemophilia. Until now, published data mainly reports in vitro pharmacodynamics and pharmacokinetics of TFPI inhibitors. Hence, in vivo effects of TFPI inhibition remain unclear, especially in haemophilia patients.

The clinical development of such molecules requires a dedicated biological monitoring. Thrombin Generation Assay (TGA) in Poor Platelets Plasma (PPP) is a good candidate since it is sensitive to Factor VIII and Factor IX deficiencies as well as to TFPI. However, TGA results are very dependent on experimental conditions (i. e. Tissue Factor and phospholipids concentrations) and the relationship between TFPI plasma level and TGA parameters has not been studied yet. This study should provide with original data on TFPI plasma levels and the effect of TFPI on thrombin generation in haemophilia patients. This should help to define the monitoring of TFPI inhibitors in Haemophilia.

DETAILED DESCRIPTION:
This study is a single-institution cohort study. Patients will be informed during their follow-up consultation. If the patient agrees to participate to this study, a non-opposition form will be signed.

If blood tests are prescribed during the consultation, the unused plasma samples that are not required to perform the prescribed analyses will be collected and anonymized in order to measure the TGA and TFPI levels.

TFPI plasmatic level and TFPI activity measurements will be performed by a quantitative ELISA assay (Total TFPI ELISA kit®, R&d Systems) and a chromogenic assay (Actichrom TFPI®, Cryopep) respectively.

TGA will be performed on a Fluoroskan® machine using 3 different levels of Tissue Factor (TF): 1, 5 and 20 pM. In order to study the relation between different levels of TFPI inhibitors and TGA parameters, TGA will also be performed by spiking blood samples with several concentrations of TFPI inhibitor. For each TGA performed, ETP (Endogenous Thrombin Potential, nM/min), peak (nM) and lagtime (min) will be analyzed.

Clinical data will be collected from the computerized patient record: date of birth, age, gender, haemophilia type (A or B) and its severity, ongoing treatments and deficient factor level.

The goal of this study is to measure the TFPI plasma level in haemophilia patients. The second objective is to assess the effects of TFPI inhibition on thrombin generation. This study should provide with original data on TFPI plasma levels and the effect of TFPI on thrombin generation in haemophilia patients. This should help to define the monitoring of TFPI inhibitors in Haemophilia.

There is no additional risk for the patient since only unused blood samples, not needed for the prescribed blood tests, will be collected.

ELIGIBILITY:
inclusion criteria :

* Men, adult (≥ 18 years old), haemophilia A or B disease (whatever the severity)
* Follow-up consultation in our center
* Blood samples collection planed during the consultation exclusion criteria :
* Children (< 18 years old), women
* No blood samples collection planed during the follow-up consultation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥ 18 years old) men haemophilia patients with follow-up consultation in our center and for whom blood tests are prescribed during the consultation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of TFPI plasma level | Day 1
  Correlation coefficient between concentration of TFPI inhibitor and parameter of thrombin generation

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France